CLINICAL TRIAL: NCT02171455
Title: Safety, Pharmacodynamics and Pharmacokinetics After Single Oral Administration of 600 mg, 750 mg and 900 mg Dabigatran Etexilate as Capsule in Healthy Subjects. A Randomised, Placebo-controlled Study, Double Blind at Each Dose Level
Brief Title: Safety, Pharmacodynamics and Pharmacokinetics After Single Oral Administration of Dabigatran Etexilate Capsule in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.60
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (3):
- Dabigatran etexilate low dose (Experimental)
  Interventions: Drug: Dabigatran etexilate low dose; Drug: Placebo
- Dabigatran etexilate medium dose (Experimental)
  Interventions: Drug: Dabigatran etexilate medium dose; Drug: Placebo
- Dabigatran etexilate high dose (Experimental)
  Interventions: Drug: Dabigatran etexilate high dose; Drug: Placebo

INTERVENTIONS:
Drug: Dabigatran etexilate low dose
  Arms: Dabigatran etexilate low dose
Drug: Dabigatran etexilate medium dose
  Arms: Dabigatran etexilate medium dose
Drug: Dabigatran etexilate high dose
  Arms: Dabigatran etexilate high dose
Drug: Placebo

SUMMARY:
To assess safety, pharmacokinetics and the effect of dabigatran on coagulation parameters prior to administration of a high dose of dabigatran etexilate in a QT study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age ≥18 and ≤55 years
3. Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Inability to comply with dietary regimen of study centre

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Frequency [N (%)] of subjects with adverse events | up to 18 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of free and total BIBR 953 ZW in plasma) | up to 72 hours after administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after administration
AUC0-∞ (area under the concentration-time curve of free and total BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after administration
λz (terminal rate constant in plasma) | up to 72 hours after administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 72 hours after administration
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours after administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 72 hours after administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 72 hours after administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 72 hours after administration